CLINICAL TRIAL: NCT04815044
Title: Experiences From Pregnancy and Post-partum Period, and Health Outcomes for Mother and Child, in Women With a History of Eating Disorders.
Brief Title: Experiences From Pregnancy and Post-partum Period in Women With a History of Eating Disorders.
Acronym: PREG_PED-t
Status: Completed | Type: Observational
Sponsor: Ostfold University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate Professor, Ostfold University College
Other Study IDs: 120532
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder; Post Partum Depression
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder; Depression, Postpartum | interventions — Pregnancy; Postpartum Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women from the PED-t study: Women who participated in the PED-t study in 2016-2018 who report previous (or in future time) pregnancy.
  Interventions: Other: Pregnancy; Other: Post-Partum

INTERVENTIONS:
Other: Pregnancy — Experiences from being pregnant when having a history of eating disorder
Other: Post-Partum — Experiences from the post-partum period when having a history of eating disorder

SUMMARY:
Women with the eating disorder bulimia nervosa (BN) have been found to have a higher risk of unplanned pregnancies than healthy women, and experience greater miscarriage, premature birth, birth complications, and postpartum depression. Other studies have found that women with eating disorders seem to find motivation to refrain from the eating disordered behavior for the sake of the fetus, but that it is highly different whether this gives sustained or only a temporary remission.

Eating disorders are rarely detected in the primary health care service, nor during pregnancy or during follow-up in fertility clinics. Meeting a health care provider in the pregnancy care service who does not know about the eating disorder or who does not understand the disease well enough, can also make the management and experience of pregnancy and weight gain extra difficult.

The aim of this study is to increase the knowledge on how women with a history of eating disorder experience their bodily changes, and how they experience the health service in pregnancy care and post-partum period.

DETAILED DESCRIPTION:
Women with the eating disorder bulimia nervosa (BN) have been found to have a higher risk of unplanned pregnancies than healthy women, and experience greater miscarriage, premature birth, birth complications, and postpartum depression. Having a disorder in which the overevaluation of the need to control body weight and food intake is pertinent, may cause a tremendous mental challenge to accept the bodily change through a pregnancy. Other studies have found that women with eating disorders seem to find motivation to refrain from the eating disordered behavior for the sake of the fetus, but that it is highly different whether this gives sustained or only a temporary remission.

Eating disorders are rarely detected in the primary health care service, nor during pregnancy or during follow-up in fertility clinics. Meeting a health care provider in the pregnancy care service who does not know about the eating disorder or who does not understand the disease well enough, can also make the management and experience of pregnancy and weight gain extra difficult.

The aim of this study is to increase the knowledge on how women with a hisory of eating disorders experience bodily changes through pregnancy, and how the pregnancy care service is experienced. The purpose of this data collection is to help design preparatory information for women with eating disorders who become pregnant, and to promote best practice guidelines for the health service in the meeting with, and follow-up of, pregnant women with a history of eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* previous participant in the PED-t project
* previous/current diagnosis of bulimia nervosa or binge eating disorder
* has accepted to take part in the long-term follow up study in the PED-t project
* has been/are pregnant

Exclusion Criteria:

* not matching the above criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Qualifying women are those who during 2016-2018 participated in the treatment project "PED-t", in which women with bulimia nervosa or binge eating disorder received PED-t or cogntive behavior therapy as treatment for their eating disorder.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Experiences of bodily changes in pregnancy and post-partum period | January 2021 - December 2026
  What are the experiences of bodily changes in pregnancy and post-partum period in women with a history of eating disorders? (semistructured interviews)
Experiences with pregnancy health care- and post-partum service | January 2021 - December 2026
  What are the experiences of pregnancy health care service in women with a history of eating disorders? (semistructured interviews)
Quality of prenatal care | January 2021 - December 2026
  Questionnaire rating (Likert scale 0, don't agree - 5, totaly agree) different aspects in the prenatal care service

SECONDARY OUTCOMES:
Current symptoms of eating disorders | January 2021 - December 2026
  Measuring current symptoms of eating disorders at time of interview. Using the eating disorder examination questionnaire by Fairburn.
Current symptoms of depression | January 2021 - December 2026
  Measuring current symptoms of depression at time of interview. Using the Beck Depression inventory.
Planning of pregnancy | January 2021 - December 2026
  Number of pregnancy that was (un)planned, and whether the female was using hormonal contraceptives at time of conception.
Help in becoming pregnant | January 2021 - December 2026
  Number of women in need of fertility assistance/treatment
Supplementation and drugs during pregnancy | January 2021 - December 2026
  Number of women who regularly consumed tobacco/were smoking, drank alcohol, or used prescribed drugs during pregnancy
Body weight during pregnancy | January 2021 - December 2026
  Change in body weight during pregnancy
Blood pressure in pregnancy | January 2021 - December 2026
  Change in blood pressure during pregnancy
Fetus heart rate | January 2021 - December 2026
  Change in fetus heart rate during pregnancy
Symphysis measure | January 2021 - December 2026
  Change in symphysis measure during pregnancy
Frequency and type of pregnancy complication | January 2021 - December 2026
  Numbers experiences different pregnancy complications (chosing from a list of alternatives: abortion, bleedings, edema, gestational diabetes, preeclampsia, pelvic pain)
Birth delivery method | January 2021 - December 2026
  Frequency of different birth delivery methods

OTHER OUTCOMES:
Exercise in pregnancy, frequency | January 2021 - December 2026
  Change in exercise frequency during pregnancy
Exercise in pregnancy, intensity | January 2021 - December 2026
  Change in exercise intensity during pregnancy
Exercise in pregnancy, activity type | January 2021 - December 2026
  Type of physical activity during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Østfold University College
Locations (1):
- Therese Fostervold Mathisen, Fredrikstad, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No
Data will be held within the research group